CLINICAL TRIAL: NCT03358433
Title: Effectiveness of Exercise in the Treatment of Depression in Older People as an Alternative to Drugs Antidepressants in Primary Care
Brief Title: Effectiveness of Exercise in the Treatment of Depression
Acronym: DEP-EXERCISE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gerencia de Atención Primaria, Albacete (Other)
Responsible Party: Principal Investigator, Jesús López-Torres Hidalgo, MD, Gerencia de Atención Primaria, Albacete
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI15/01486
Record Dates: First submitted 2017-11-25; First posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Depression; Primary Care; Exercise
MeSH Terms: conditions — Depression; Motor Activity | interventions — Exercise; Antidepressive Agents

ARMS (2):
- Exercise (Experimental)
  Interventions: Other: Exercise
- Antidepressants (Active Comparator)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise
  Other Names: Antidepressants

SUMMARY:
The main objective is to test the non-inferiority of supervised exercise versus antidepressant treatment in reducing depressive symptoms in patients with clinical criteria for depression (according to ICD 10) over a period of 6 months follow-up.

DETAILED DESCRIPTION:
This is a randomized clinical trial in primary care in which a total of 312 patients over 65 years with clinically significant depression will be randomly assigned to an exercise program supervised or receive treatment with antidepressant drugs commonly used in clinical practice. At baseline physical fitness of the participants will be checked, and assessments will be made after 15 days and 1, 3 and 6 months. The supervised exercise program will consist of 2 sessions per week in groups of 10-12 patients over a 6 month period in which a sports instructor will train patients to perform at least 30 minutes of regular, moderate-intensity activity with a frequency almost daily, including aerobic exercise and strength training, flexibility and balance. In both groups will be evaluated periodically, among other variables, the state of depressive symptoms, level of physical activity, self-rated health, occurrence of adverse effects and adherence to exercise program or antidepressant treatment. The main outcome measure is the reduction of the baseline score on the scales of depressive symptoms (Montgomery-Asberg Depression Rating Scale and Geriatric Depression Scale).

ELIGIBILITY:
Inclusion Criteria:

* People with depression

Exclusion Criteria:

* Contraindication to exercise

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2016-06-01 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement in depressive symptoms | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jesús López-Torres Hidalgo, MD, Principal Investigator — Centro de Salud Zona VIII de Albacete (Spain)
Locations (2):
- Spain (2):
  - Jesús López-Torres Hidalgo, Albacete
  - Albacete

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hidalgo JL, Sotos JR; DEP-EXERCISE Group. Effectiveness of Physical Exercise in Older Adults With Mild to Moderate Depression. Ann Fam Med. 2021 Jul-Aug;19(4):302-309. doi: 10.1370/afm.2670. PMID 34264835
- [Derived] Lopez-Torres Hidalgo J; DEP-EXERCISE Group. Effectiveness of physical exercise in the treatment of depression in older adults as an alternative to antidepressant drugs in primary care. BMC Psychiatry. 2019 Jan 14;19(1):21. doi: 10.1186/s12888-018-1982-6. PMID 30642326